CLINICAL TRIAL: NCT03822949
Title: Bright Light Exposure in Patients Undergoing Non-cardiac Elective Surgery
Brief Title: Bright Light Exposure in Surgical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-0904; R01HL122472 (NIH)
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Ischemia; Critical Illness; Endothelial Dysfunction
MeSH Terms: conditions — Myocardial Ischemia; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Experimental: Exposed to Day light (Experimental): Patients undergoing primary sternotomy cardiac surgery: Patients will be enrolled 10 to 1 days prior to surgery and will receive an intense (bright light, Square One Wake Up Light NatureBright 10,000 LUX) box. The patient will start using the light box prior to surgery every morning from 8.30 to 9.00 AM. Blood /buccal swabs will be collected on the day of enrollment (10 to 1 days prior to surgery) between 7 and 10 AM without any light therapy and on the day of surgery between 7 and 10 AM before anesthesia induction after one week of light therapy.
  Interventions: Device: Day Light
- Sham Comparator: Exposed to Room light (Placebo Comparator): Patients undergoing primary sternotomy cardiac surgery: Patients will be enrolled 10 to 1 days prior to surgery and will receive a placebo/control device (dim/night light box). The patient will start using the light box 7 days prior to surgery every morning from 8.30 to 9.00 AM. Blood /buccal swabs will be collected on the day of enrollment (10 to 1 days prior to surgery) between 7 and 10 AM without any light therapy and on the day of surgery between 7 and 10 AM before anesthesia induction after one week of placebo therapy.
  Interventions: Device: Placebo light
- Experimental: ICU Exposed to Day light (Experimental): Patients undergoing trauma or elective surgery with ICU admission: Light therapy will consist of 30 minutes intense light each morning for 5-10 days. Blood will be drawn before sunrise and after light therapy. Light therapy will be performed by a study nurse to ensure proper use. In addition, endothelial function and activity will be measured using the noninvasive Endo-pat and ActiWatch device. The patient will need to keep the box as close as possible to their eyes and not walk away during the treatment period. This will be facilities by a study nurse.
  Interventions: Device: ICU Intense Light
- Sham Comparator: ICU Exposed to Room light (Placebo Comparator): Patients undergoing trauma or elective surgery with ICU admission: Light therapy will consist of 30 minutes using a placebo/control device (dim/night light box) each morning for 5-10 days. Blood will be drawn before sunrise and after light therapy. Light therapy will be performed by a study nurse to ensure proper use. In addition, endothelial function and activity will be measured using the noninvasive Endo-pat and ActiWatch device.
  Interventions: Device: ICU Placebo light

INTERVENTIONS:
Device: Day Light — Patients are exposed to daylight for up to 10 days prior to surgery
  Arms: Experimental: Exposed to Day light
Device: Placebo light — Patients are exposed to placebo light for up to 10 days prior to surgery
  Arms: Sham Comparator: Exposed to Room light
Device: ICU Intense Light — ICU Patients are exposed to daylight for up to 10 days after surgery
  Arms: Experimental: ICU Exposed to Day light
Device: ICU Placebo light — ICU Patients are exposed to placebo light for up to 10 days after surgery
  Arms: Sham Comparator: ICU Exposed to Room light

SUMMARY:
1. Elucidate the influence of intense light therapy pretreatment in patients undergoing cardiac surgery. We hypothesize that intense light exposure is associated with the peripheral stabilization of Per2 in human buccal swabs and plasma samples before surgery and with a decrease of Troponin I levels after surgery. In addition, we hypothesize that light therapy leads to Per2 dependent metabolic optimization in the human cardiac tissue. Therefore, a small piece of human heart tissue from the right atrium will be collected during cardiac cannulation, which will be otherwise discarded.
2. Critical illness (being in the intensive care unit) results in circadian malfunction and vessels not working. Vessel function is controlled by the body's circadian clock. Intense light boosts the circadian clock and the vessel function in animal studies. Vessels not working well in critical ill patients results in a myriad of severe diseases (delirium, stroke, heart attack, organ damage etc). Thus we will test if intense light can be used to boost the circadian clock and the associated vessel function in critical ill patients.

DETAILED DESCRIPTION:
PER2 transcript and protein levels in patients undergoing cardiac surgery following intense light therapy utilizing blood samples, buccal swaps and right atrial myocardium. In addition, we will examine the correlation of PER2 levels and PER2 related metabolism and perform a whole genome microarray screen from the collected tissue/blood samples.

Patients will be enrolled 10 to 1 days prior to surgery and will either receive an intense (bright light) box or a placebo/control device (dim/night light box). The patient will start using the light box 7 days prior to surgery every morning from 8.30 to 9.00 AM. The patient will need to keep the box as close as possible to their eyes and not walk away during the treatment period.

1. Blood /buccal swabs will be collected on the day of enrollment (10-1 days prior to surgery) between 7 and 10 AM without any light therapy and on the day of surgery between 7 and 10 AM before anesthesia induction after one week of light/placebo therapy.

   A small piece of the right atrial myocardium (which stems from cardiac cannulation and is otherwise discarded) will be put in liquid nitrogen in the OR and stored for further analysis.

   In addition, we will draw a blood sample 72 hrs. after surgery and determine Troponin I levels.

   Investigating this patient population will give the necessary evidence if light could also be effective in a perioperative setting to prevent or decrease damage to the myocardium during high risk cardiac surgery. In addition, it will help us understand if light could be used in general to prevent or treat heart ischemia.
2. We will use our light boxes for 30 minutes in ICU care patients on the first morning after admission from 8.30 to 9.00 AM. Before light therapy/sunrise and immediately after light therapy, a blood sample is drawn. These samples will be analyzed for melatonin levels. We have demonstrated that effective intense blue intense light therapy significantly suppresses melatonin plasma levels in health human volunteers which is the desired outcome of light therapy. We also have shown that light exposure via windows does not achieve such a result. Light therapy will be continued for up to 10 days, and blood samples are drawn each morning before sunrise and after light therapy. In patients that are sedated and have their eyes closed, eyes will be opened manually and lubricated before light therapy is initiated. The sample size will be n=40 (10 light treatment 5 days, 10 light treatment 10 days and 10 standard room light treatment 5 and 10 days). Additional readouts from plasma sample will be triglyceride and ANGPTL4 levels as we have already shown that intense light significantly downregulates triglycerides in healthy volunteers. Further, we recently discovered ANGPTL4 as major light dependent protein. ANGPTL4 is a key regulator of triglycerides and of endothelial function in humans and triglyceride levels are also indicative of endothelial function. This approach will allow us to evaluate the effectiveness of our light therapy approach and will further give insight into light elicited endothelial mechanisms in humans.

To further study endothelial function, we will use the Endo_PAT device (Itamar Medical Ltd, Franklin, MA) which has been shown to reliably detect endothelial dysfunction and alterations in critical ill patients. This device has been shown to even work when patients who are on vasopressor therapy. This device is noninvasive and works like an SpO2 monitor with built in cuff pressure measurement.

Finally, we will use Actigraphy (Actiwatch, Phillips) to analyze circadian patterns and associated changes following light therapy. We already have purchased FDA approved Actigraphy devices and shown that intense light strengthens the circadian rhythms in healthy volunteers. Watches will be around the wrist for the duration of the light therapy and are noninvasive.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary sternotomy cardiac surgery
* Subjects in the range of 18 - 90 years old .
* Patient need to be in sinus rhythm at the time of surgery.

Exclusion Criteria:

* patients <18 or >90 years old
* participation in other clinical trials within the previous 30 days
* pregnancy
* neurological conditions that could impair weaning from ventilator support
* significant CNS disorders or comorbid irreversible conditions with a six-month mortality rate more than 50 percent
* prisoners, or subjects with altered capabilities to make decision will be enrolled
* medical history of type 2 diabetes
* patients with atrial fibrillation or use of class III anti-arhythmic drug
* patients with a left ventricle ejection fraction < 40%
* patient in emergency condition

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-07-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change of Period 2 (Per2) protein levels | 1-10 days
  Measure of Per2 protein levels related to daylight exposure vs. room light exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Eckle, MD, PhD, Principal Investigator — UC Denver
Locations (1):
- University of Colorado Denver | Anschutz Medical Campus, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartman CM, Oyama Y, Eckle T. Daytime variations in perioperative myocardial injury. Lancet. 2018 May 26;391(10135):2104. doi: 10.1016/S0140-6736(18)30797-9. Epub 2018 May 24. No abstract available. PMID 29856340
- [Background] Oyama Y, Bartman CM, Gile J, Eckle T. Circadian MicroRNAs in Cardioprotection. Curr Pharm Des. 2017;23(25):3723-3730. doi: 10.2174/1381612823666170707165319. PMID 28699517
- [Background] Bonney S, Hughes K, Harter PN, Mittelbronn M, Walker L, Eckle T. Cardiac period 2 in myocardial ischemia: clinical implications of a light dependent protein. Int J Biochem Cell Biol. 2013 Mar;45(3):667-71. doi: 10.1016/j.biocel.2012.12.022. Epub 2013 Jan 3. PMID 23291353
- [Result] Oyama Y, Bartman CM, Gile J, Sehrt D, Eckle T. The Circadian PER2 Enhancer Nobiletin Reverses the Deleterious Effects of Midazolam in Myocardial Ischemia and Reperfusion Injury. Curr Pharm Des. 2018;24(28):3376-3383. doi: 10.2174/1381612824666180924102530. PMID 30246635
- [Result] Bartman CM, Oyama Y, Brodsky K, Khailova L, Walker L, Koeppen M, Eckle T. Intense light-elicited upregulation of miR-21 facilitates glycolysis and cardioprotection through Per2-dependent mechanisms. PLoS One. 2017 Apr 27;12(4):e0176243. doi: 10.1371/journal.pone.0176243. eCollection 2017. PMID 28448534
- [Result] Bonney S, Kominsky D, Brodsky K, Eltzschig H, Walker L, Eckle T. Cardiac Per2 functions as novel link between fatty acid metabolism and myocardial inflammation during ischemia and reperfusion injury of the heart. PLoS One. 2013 Aug 20;8(8):e71493. doi: 10.1371/journal.pone.0071493. eCollection 2013. PMID 23977055
- [Result] Eckle T, Hartmann K, Bonney S, Reithel S, Mittelbronn M, Walker LA, Lowes BD, Han J, Borchers CH, Buttrick PM, Kominsky DJ, Colgan SP, Eltzschig HK. Adora2b-elicited Per2 stabilization promotes a HIF-dependent metabolic switch crucial for myocardial adaptation to ischemia. Nat Med. 2012 Apr 15;18(5):774-82. doi: 10.1038/nm.2728. PMID 22504483